CLINICAL TRIAL: NCT00727376
Title: Clinical Evaluation of Polyflex Stenting in Esophageal Cancer Patients Undergoing Chemotherapy and/or Radiation Therapy
Brief Title: Evaluation of Polyflex Stenting in Esophageal Cancer Patients
Status: Completed | Type: Observational
Sponsor: University of Louisville (Other)
Responsible Party: Principal Investigator, Robert C. Martin, Professor, University of Louisville
Other Study IDs: 08-0132
Record Dates: First submitted 2008-07-30; First posted 2008-08-04 (Estimated); Last update posted 2020-08-03 (Actual); Status verified 2018-03

CONDITIONS: Esophageal Cancer
Keywords: esophageal; stenting
MeSH Terms: conditions — Esophageal Neoplasms

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No

GROUPS / COHORTS (1):
- Observation: Esophageal cancer patients

SUMMARY:
To evaluate the effectiveness of an esophageal stent as a way to maintain nutrition during radiation and/or chemotherapy treatment.

ELIGIBILITY:
Inclusion Criteria:

* 18 years of age and older
* Willing and able to provide informed consent
* Willing to comply with follow-up requirements
* Biopsy-confirmed esophageal cancer (adenocarcinoma or squamous cell carcinoma) in mid or distal esophagus (clinical stage 3 or less)
* Indicated for chemotherapy and/or radiation therapy
* Ability to dilate stricture to 15mm diameter at extent of disease evaluation
* Placement of at least 18 x 23mm diameter and 120mm length PolyFlex stent

Exclusion Criteria:

* Patients contraindicated for endoscopy
* Patients with prior esophageal stent placements
* Advance stage of disease, greater than T3 tumor or M1 disease

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Esophageal cancer patients who have elected to have a stent placed.
Sampling Method: Non-Probability Sample
Enrollment: 26 (Actual)
Dates: Start 2008-03; Primary Completion 2011-02 (Actual); Study Completion 2011-02 (Actual)

PRIMARY OUTCOMES:
Clinical benefit of the Polyflex Esophageal Stent as a means to maintain oral nutrition during chemotherapy and/or radiation | 8 - 10 weeks

CONTACTS AND LOCATIONS:
Overall Officials: Robert Martin, MD, Principal Investigator — University of Louisville
Locations (1):
- University of Louisville, Louisville, Kentucky, United States

REFERENCES:
- [Derived] Martin RC 2nd, Cannon RM, Brown RE, Ellis SF, Williams S, Scoggins CR, Abbas AE. Evaluation of quality of life following placement of self-expanding plastic stents as a bridge to surgery in patients receiving neoadjuvant therapy for esophageal cancer. Oncologist. 2014 Mar;19(3):259-65. doi: 10.1634/theoncologist.2013-0344. Epub 2014 Feb 24. PMID 24567281
- [Derived] Brown RE, Abbas AE, Ellis S, Williams S, Scoggins CR, McMasters KM, Martin RC 2nd. A prospective phase II evaluation of esophageal stenting for neoadjuvant therapy for esophageal cancer: optimal performance and surgical safety. J Am Coll Surg. 2011 Apr;212(4):582-8; discussion 588-9. doi: 10.1016/j.jamcollsurg.2010.12.026. PMID 21463793